CLINICAL TRIAL: NCT00389584
Title: Phase I/II Study of Irinotecan and Whole Brain Radiation Therapy in Patients With Brain Metastases From Solid Tumors
Brief Title: Irinotecan and Whole-Brain Radiation Therapy in Treating Patients With Brain Metastases From Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Allan Y. Chen, MD, PhD, Assistant Professor (no longer at UC Davis); not to be confused with Allen M. Chen, MD
Purpose: Treatment
Other Study IDs: CDR0000506074; UCDCC-132; UCDCC-200210643-5; PFIZER-Z1001692
Record Dates: First submitted 2006-10-18; First posted 2006-10-19 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Brain and Central Nervous System Tumors; Cognitive/Functional Effects; Long-term Effects Secondary to Cancer Therapy in Adults; Long-term Effects Secondary to Cancer Therapy in Children; Poor Performance Status; Unspecified Adult Solid Tumor, Protocol Specific; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: cognitive/functional effects; poor performance status; long-term effects secondary to cancer therapy in adults; long-term effects secondary to cancer therapy in children; adult tumors metastatic to brain; unspecified adult solid tumor, protocol specific; unspecified childhood solid tumor, protocol specific
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms | interventions — Irinotecan; Mental Status and Dementia Tests; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: irinotecan hydrochloride
Procedure: cognitive assessment
Procedure: management of therapy complications
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as irinotecan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Irinotecan may make tumor cells more sensitive to radiation therapy. Giving irinotecan together with whole-brain radiation therapy may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of irinotecan when given together with whole-brain radiation therapy and to see how well they work in treating patients with brain metastases from solid tumors. (The study of side effects and best dose has ended as of 4/15/05)

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of irinotecan hydrochloride administered concurrently with whole-brain radiotherapy in patients with brain metastases from solid tumors. (Phase I) (Phase I closed to accrual as of 4/15/05)
* Determine the toxicity of this regimen in these patients. (Phase I) (Phase I closed to accrual as of 4/15/05)
* Determine the overall survival of patients treated with this regimen. (Phase II)

Secondary

* Assess the neurocognitive function of these patients by Mini-Mental Status Examination. (Phase II)

OUTLINE: This is a phase I, dose-escalation study of irinotecan hydrochloride (phase I closed to accrual as of 4/15/05) followed by a phase II study. Patients enrolled in phase II are stratified according to cognitive dysfunction (yes vs no).

* Phase I (closed to accrual as of 4/15/05): Patients undergo whole-brain radiotherapy (WBRT) once daily, 5 days a week, for 3 weeks (15 fractions). Patients also receive irinotecan hydrochloride IV over 90 minutes on days 1, 8, and 15.

Cohorts of 3-6 patients receive escalating doses of irinotecan hydrochloride until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

* Phase II (for patients enrolled after 4/15/05): Patients receive irinotecan hydrochloride at the MTD and undergo concurrent WBRT as in phase I.

Patients complete the Mini-Mental Status Examination to assess neurocognitive function at baseline, on the last day of radiotherapy, and periodically after completion of study therapy.

After completion of study therapy, patients are followed monthly for 3 months, at 6 months, and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 51 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of brain metastasis from a histologically confirmed solid tumor, meeting the following criteria:

  * Must have histologic proof of original malignancy
  * No germ cell tumor metastasis
  * Biopsy-proven brain metastasis preferred when clinical history and radiographic findings are equivocal
* At least 1 unidimensionally measurable lesion ≥ 50 mm by head contrast CT scan and/or brain MRI
* Patients enrolled in the phase II portion of the study must meet the following Radiation Therapy Oncology Group Recursive Partitioning Analysis staging criteria for brain metastases:

  * Class II classification

    * Zubrod performance status 0-1 AND any of the following:

      * Age > 65 years
      * Extracranial metastasis
      * Uncontrolled primary malignancy

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-1
* Life expectancy ≥ 3 months
* Able to participate in the Mini-Mental Status Examination
* WBC ≥ 3,000/mm³
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin ≤ 1.5 mg/dL
* AST ≤ 2.5 times upper limit of normal (ULN) (5 times ULN if liver metastases are present)
* Hemoglobin ≥ 9.0 g/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No concurrent medical disease that, in the investigator's opinion, would preclude study participation

PRIOR CONCURRENT THERAPY:

* More than 21 days since prior chemotherapy
* No prior whole-brain radiotherapy
* No prior DNA topoisomerase I drugs (e.g., irinotecan hydrochloride, topotecan hydrochloride)
* At least 4 days since prior and no concurrent known CYP3A4 inducers, including any of the following:

  * Phenytoin
  * Carbamazepine
  * Phenobarbital
  * Hypericum perforatum (St. John's wort)

Ages: 1 Year to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2002-12; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose and toxicity as assessed by NCI CTC v2.0 (Phase I) (Phase I closed to accrual as of 4/15/05)
Overall survival (Phase II)

SECONDARY OUTCOMES:
Neurocognitive deterioration as assessed by Mini-Mental Status Examination (Phase II)
Time to cognitive failure as assessed by Kaplan-Meier (Phase II)

CONTACTS AND LOCATIONS:
Overall Officials: Allan Y. Chen, MD, PhD, Study Chair — University of California, Davis
Locations (1):
- University of California Davis Cancer Center, Sacramento, California, United States